CLINICAL TRIAL: NCT02350621
Title: Cervical Foraminal Stenosis and Radiculopathy - Anterior Cervical Discectomy and Fusion (ACDF) Versus Minimal Invasive Posterior Cervical Foraminotomy miPCF).
Brief Title: Cervical Foraminal Stenosis and Radiculopathy - ACDF Versus Minimal Invasive Posterior Cervical Foraminotomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stockholm Spine Center AB (Other)
Responsible Party: Principal Investigator, Andreas Selander, MD, Stockholm Spine Center AB
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/1150-31/2
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Radiculopathy
Keywords: cervical foraminal stenosis minimal invasive foraminotomy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACDF (Active Comparator): Anterior Cervical Discectomy and Fusion
  Interventions: Procedure: ACDF
- miPCF (Active Comparator): minimal invasive Posterior Cervical Foraminotomy
  Interventions: Procedure: minimal invasive Posterior Cervical Foraminotomy

INTERVENTIONS:
Procedure: ACDF
  Arms: ACDF
Procedure: minimal invasive Posterior Cervical Foraminotomy
  Arms: miPCF

SUMMARY:
A prospective randomized clinical trial. Cervical spondylotic foraminal stenosis with radiculopahty. Comparison results between 2 treatment options: ACDF and minimal invasive posterior cervical foraminiotomy.

80 patients to be followed for 2 years. Parameters to study: NDI, VAS, EQ-5D, complications, health economics, recurrens of stenosis, movement of facet joints pre- and postoperatively (foraminotomy group).

ELIGIBILITY:
Inclusion Criteria:

* Cervical radiculopathy on 1 or 2 levels correlated on MRI and CT Arm pain more than 30 (VAS). Duration more than 3 months.

Exclusion Criteria:

* Myelopathy. Soft disc hernia. Previous neck surgery. Tumors, infection, WAD, trauma, generalized pain syndrome.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Tycho Tullberg, MD, PhD, Study Chair — Stockholm Spine Center